CLINICAL TRIAL: NCT00215059
Title: Measurement of Angiogenic Related Growth Factors in Urine and Blood From Patients With Multivessel Pulmonary Vein Stenosis
Brief Title: Measurement of Angiogenic Related Growth Factors in Urine and Blood From Patients With Pulmonary Vein Stenosis
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Boston Children's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Mark Kieran, Children's Hospital Boston
Other Study IDs: CH X00-09-050
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Multivessel Pulmonary Vein Stenosis
Keywords: angiogenic related growth factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, single center, descriptive study in 14 infants/children with multivessel pulmonary vein stenosis stratified for patients with or without underlying cardiac disease.

Group 1: Patients without additional structural heart disease and multivessel pulmonary vein stenosis.

Group 2: Patients with additional structural heart disease and multivessel pulmonary vein stenosis.

DETAILED DESCRIPTION:
Patients identified at the time of presentation to their cardiologist will be asked to provide a urine sample for analysis. If blood is being drawn for other clinical tests, an extra vial of blood will be collected for measurement of bFGF, VEGF, angiopoietin 1&2 and ephrin. At the time of blood draws, approximately 4 cc's of heparin blood will be obtained and processed as detailed below. Blood and/or urine samples will be coordinated through the data manager and will be performed only when blood is being obtained for other reasons. Initially, blood samples will be sent to Lab Control, spun down, and the plasma isolated. Plasma will be coded, then frozen at -200C in the research lab. Urine samples will be aliquoted into vials and stored at -20 until further analysis.

All patient information will be kept confidential. Individual results will not be provided to patients. Identifiers to patient information will be maintained. No identifying patient information will be used in publications that might result from these studies. Information to be collected by the data manager will include age, sex, date of diagnosis and interventions.

The specific aim is to assess angiogenic growth factor concentrations in urine and blood from patients with both congenital and acquired multivessel pulmonary vein stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis can be based on clinical and radiographic grounds or at the time of biopsy or prior surgical procedures. The diagnosis must be consistent with multivessel pulmonary stenosis.
* There must be evidence of severe pulmonary vein stenosis in at least two pulmonary veins.
* Must give written informed consent according to institutional guidelines

Exclusion Criteria:

* Mechanism of pulmonary venous obstruction due to obvious anatomic cause, such as extrinsic compression

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with pulmonary vein stenosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2000-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Kieran, MD,PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts